CLINICAL TRIAL: NCT00837902
Title: Genetic Determinants of Response to Beta Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine,. Professor of Pharmacology, Assistant Director of the Division of Clinical Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 081267; P01HL056693 (NIH); U01HL065962 (NIH); 1UL1RR024975 (NIH)
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Atenolol; Exercise; Genotype; Healthy volunteers
MeSH Terms: conditions — Motor Activity | interventions — Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atenolol (Experimental): There is only 1 arm to this study. Intervention: All participants received atenolol. Genotyping for GRK5 was performed to identify if participants were GLN/GLN, GLN/LEU, or LEU/LEU.
  Heart rates were measured at rest, and as participants performed graded incremental exercise on a supine bicycle ergometer (at 25, 50, and 75 W for 2 minutes each) twice, once before and once 2.5 hours after taking 25 mg of atenolol.
  Interventions: Drug: Atenolol (β-blocker)

INTERVENTIONS:
Drug: Atenolol (β-blocker) — 25 mg tablet
  Other Names: generic atenolol is being used, so not applicable

SUMMARY:
The overall goal of this project is to determine the genetic factors contributing to interindividual differences in response to beta-blockade.

DETAILED DESCRIPTION:
The Aim is to define the contribution of genetic variation to the interindividual variability in response to β-blockade. The rationale for the study is as follows: Beta-blockers prevent the activation of β-ARs and thus form the cornerstone of treatment of pathological states such as congestive heart failure and coronary artery disease. Functional polymorphisms in cardiac beta-receptors have been shown to determine response to β-blocker therapy. A physiologic stimulus such as exercise causes sympathetic stimulation and activation of the cardiac β-ARs and genotypic differences in response to β-blockers are magnified under states of heightened sympathetic activity. Thus, in addition to measuring the response to β-blockers at rest, we will also determine the response to β-blockade after sub-maximal exercise on a supine bicycle ergometer. Genetic variations that may alter sensitivity to a beta blocker will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give written informed consent and be able to adhere to diet and study schedules.
* Subjects must be free of any clinically significant disease that requires a physician's care and/or would interfere with the study evaluations.
* Subjects must have a clinically acceptable physical examination and ECG.
* Laboratory tests (CBC, blood chemistries, and urinalysis) must be within clinically acceptable limits.

Exclusion Criteria:

* Any subject who has taken any prescription or over-the-counter drugs, other than oral contraception if female, within one week prior to study drug administration.
* Subjects who are presently, or were formerly, narcotic addicts or alcoholics.
* Active smokers.
* Subjects who have a clinically significant allergy/intolerance to atenolol.
* Females with a positive serum/urine pregnancy test at screening.
* Females who are nursing.
* Subjects with complete heart block/ any other significant cardiovascular disease.
* Subjects with a history of asthma symptoms or medication for it within last 10 years.
* Subjects who have a systolic blood pressure < 90 mm Hg or diastolic blood pressure < 50 mm Hg or heart rate < 50/min at the screening visit or on the baseline pre drug values on the study day.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Stein, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Kurnik D, Cunningham AJ, Sofowora GG, Kohli U, Li C, Friedman EA, Muszkat M, Menon UB, Wood AJ, Stein CM. GRK5 Gln41Leu polymorphism is not associated with sensitivity to beta(1)-adrenergic blockade in humans. Pharmacogenomics. 2009 Oct;10(10):1581-7. doi: 10.2217/pgs.09.92. PMID 19842931

RESULTS

PARTICIPANT FLOW:
Groups:
- White Participants--Atenolol: Unrelated white American subjects
- Black Participants-Atenolol: Unrelated black American subjects
Period: Overall Study
Arm/Group | White Participants--Atenolol | Black Participants-Atenolol
Started | 85 | 69
Completed | 85 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- White Participants--Atenolol; Black Participants-Atenolol: Unrelated black and white American subjects were eligible to participate if they were between 18 and 50 years old and had no clinically significant abnormality based on medical history, physical exam, electrocardiogram and routine laboratory testing. Subjects were free of medications for at least 1 week. They also received an alcohol and caffeine free diet for 6 days prior to the study.
- Total: Total of all reporting groups
Arm/Group | White Participants--Atenolol | Black Participants-Atenolol | Total
Number analyzed (Participants) | 85 | 69 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (6.4) | 25.9 (6) | 26.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 87
  Male | 45 | 22 | 67
Region of Enrollment [Number; unit: participants]
  United States | 85 | 69 | 154
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 109.9 (11.4) | 112.5 (12.1) | 111.1 (11.8)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 64.0 (6.8) | 66.2 (7.5) | 65.0 (7.1)
GRK5 Genotype [Count of Participants; unit: Participants]
  GLN/GLN | 85 | 29 | 114
  GLN/LEU | 0 | 35 | 35
  LEU/LEU | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Heart Rate
Description: Reduction in heart rate based upon genotype while exercising. Participants exercised on a recumbent bike for 2 minutes at 25W, 2 minutes at 50W, and 2 minutes at 75W twice, once before taking atenolol, and once 2.5 hours after oral administration of 25 mg of atenolol. Data points represent unadjusted mean reduction in heart rate in the 3 genotype groups.
Time Frame: 2 exercise periods of 6 minutes each. 6 minutes of exercise before taking atenolol, and 6 minutes of exercise starting 2.5 hours after taking 25 mg of atenolol (2.5 hours + 6 minutes)
Population: There are 3 genotypes for GRK5, GLN/GLN, GLN/LEU, and LEU/LEU. A priori analysis plan was to compare reduction in heart rate among the 3 genotypes..
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- GLN/GLN: One of 3 genotypes for GRK5, GLN/GLN
- GLN/LEU: One of 3 genotypes for GRK5, GLN/LEU
- LEU/LEU: One of 3 genotypes for GRK5, LEU/LEU.
Arm/Group | GLN/GLN | GLN/LEU | LEU/LEU
Number analyzed (Participants) | 114 | 35 | 5
beats per minute
  0, baseline | 7.9 (7) | 6 (5.9) | 3.3 (5.4)
  2 minutes from baseline, 2 minutes exercise at 25W | 9.6 (8.2) | 8.4 (7.7) | 7.4 (4.4)
  4 minutes from baseline, 2 minutes exercise at 50W | 11.7 (7) | 10.9 (7.2) | 9.1 (3.4)
  6 minutes from baseline, 2 minutes exercise at 75W | 14 (8) | 12.4 (9.1) | 10 (6.1)

ADVERSE EVENTS:
Time Frame: 7 days. Participants were placed on an alcohol and caffeine free diet for 6 days prior to the study, which provided 150 mmol of sodium, 70mmol of potassium, and 600 mmol of calcium daily, and the study day.
Description: no adverse events
Arm/Group | White Participants--Atenolol | Black Participants-Atenolol
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/69
Other Adverse Events (participants affected / at risk) | 0/85 | 0/69

LIMITATIONS AND CAVEATS:
We cannot extrapolate our results to subjects substantially different from our study group, such as elderly subjects, cardiac patients, or patients on on chronic beta-blocker therapy, or disease states such as heart failure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No